CLINICAL TRIAL: NCT00307086
Title: An Evaluation of Bortezomib (VelcadeR ) Followed by High-Dose Melphalan and Bortezomib (VelcadeR) as Conditioning Regimen for Tandem Peripheral Blood Stem Cell Transplants in Patients With Primary Refractory Multiple Myeloma and Plasma Cell Leukemia
Brief Title: Bortezomib Followed by High-Dose Melphalan and Bortezomib as Conditioning Regimen for Tandem Stem Cell Transplants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14184; X05174
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Results first posted 2013-10-24 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2013-08

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell | interventions — Bortezomib; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous PBSCT (Other): bortezomib in combination with high-dose melphalan as a conditioning regimen for autologous peripheral blood stem cell transplant (PBSCT)
  Interventions: Drug: Bortezomib; Drug: Melphalan; Procedure: PBSCT

INTERVENTIONS:
Drug: Bortezomib — the maximum tolerated dose (MTD) of bortezomib in combination with high-dose melphalan as a conditioning regimen for autologous stem cell transplant
  Other Names: Velcade
Drug: Melphalan — Day -4 melphalan 100 mg/m2 intravenously over 30 minutes, Day -3 melphalan 100 mg/m2 intravenously over 30 minutes
  Other Names: Alkeran(R)
Procedure: PBSCT — PBSCT #1 Day 0 PBSCT #2 Day 0 (approx 90 days =/- 15 days after PBSCT #1)
  Other Names: peripheral blood stem cell transplant (PBSCT)

SUMMARY:
The primary objectives of this study are to:

* To determine the maximum tolerated dose (MTD) of bortezomib in combination with high-dose melphalan as a conditioning regimen.
* To determine the safety, tolerability, and response rates of bortezomib given in combination with high-dose melphalan, as a conditioning regimen, for tandem transplants in patients with primary refractory multiple myeloma or plasma cell leukemia.

The secondary objectives of this study are to:

* To determine gene expression profiles (pharmacogenomics) and perform RTPCR for Fanconi anemia pathway genes, prior to and after treatment with bortezomib, in patients with primary refractory multiple myeloma and plasma cell leukemia and correlate profiles with responses to treatment.
* To determine the time to disease progression and overall survival in patients with primary refractory multiple myeloma and plasma cell leukemia treated with bortezomib followed by tandem autologous transplantation
* To determine the response rates of 2 cycles of bortezomib in patients with primary refractory multiple myeloma or plasma cell leukemia

DETAILED DESCRIPTION:
Patients with primary refractory multiple myeloma or plasma cell leukemia either newly diagnosed or previously treated will receive 2-cycles of standard dose bortezomib followed by high-dose melphalan and bortezomib as a conditioning regimen prior to a tandem autologous peripheral blood stem cell transplantation (PBSCT). Following treatment with two cycles of standard dose bortezomib, sequential cohorts of patients will be given escalating bortezomib doses combined with standard and constant conditioning regimen doses of melphalan. Once the MTD of bortezomib is reached, that dose will be administered in combination with melphalan as conditioning prior to PBSCT.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male agrees to use an acceptable method for contraception for the duration of the study.
* Multiple Myeloma Criteria:
* Patients with primary refractory disease (those failing to achieve at least a partial response, as defined by the Bladé multiple myeloma response criteria, after first-line (induction) therapy). A partial response will be defined as the following: ≥50% reduction in the level of the serum monoclonal paraprotein, maintained for a minimum of 6 weeks, Reduction in 24-hour urinary light chain excretion either by ≥ 90% or to < 200 mg, maintained for a minimum of 6 weeks. For patients with non-secretory myeloma only, ≥ 50% reduction in plasma cells in a bone marrow aspirate and biopsy, maintained for a minimum of 6 weeks, ≥ 50% reduction in the size of soft tissue plasmacytomas (by radiography or physical examination). No increase in the size or number of lytic bone lesions (development of a compression fracture does not exclude response).
* Patients with plasma cell leukemia, either newly diagnosed or previously treated.
* Patients greater than or equal to 18 years of age are eligible.
* Patients must have a histologically confirmed diagnosis by a pathologic review at the H. Lee Moffitt Cancer Center and Research Institute.
* Patients must have undergone a complete psychosocial evaluation and have been considered capable of compliance.

Exclusion Criteria:

* Patient has a platelet count of <30× 10^9/L within 14 days before enrollment.
* Patient has an absolute neutrophil count of <1.0 × 10^9/L within 14 days before enrollment.
* Patient has a serum creatinine of greater than 2.0 mg/dL OR a creatinine clearance of less than 40 ml/minute within 14 days before enrollment. Creatinine clearance can be measured or calculated.
* Has >Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for postmenopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients with a DLCO less than 50% (adjusted) of normal or with symptomatic obstructive or restrictive lung disease are ineligible.
* Patients with renal dysfunction secondary to multiple myeloma may be enrolled at the discretion of the principal investigator. However, patients on hemodialysis or peritoneal dialysis are ineligible.
* Patients with a total bilirubin greater than 2.0 mg/dL and SGOT or SGPT greater than two and a half times normal (unless due to primary malignancy), or a history of severe hepatic dysfunction are ineligible.
* Patients with active infections are ineligible.
* Patients who are HIV positive are ineligible.
* Patients with active leptomeningeal involvement are ineligible. Patients with a history of previous CSF tumor involvement without symptoms or signs are eligible provided the CSF is now free of disease on lumbar puncture, and MRI of the brain shows no tumor involvement. Patients with severe symptomatic central nervous system (CNS) disease of any etiology are ineligible.
* Patients with uncontrolled insulin-dependent diabetes mellitus or uncompensated major thyroid or adrenal dysfunction are ineligible.
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 2 are ineligible.
* Patients with an ECOG performance status of 2 to 3, secondary to bone pain, may be enrolled at the discretion of the institutional investigator(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Todd Alekshun, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: H Lee Moffitt Cancer Center & Research Institute website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from the Blood and Marrow Transplant (BMT) program at H. Lee Moffitt Cancer Center.
Groups:
- Autologous PBSCT: bortezomib in combination with high-dose melphalan as a conditioning regimen for autologous peripheral blood stem cell transplant
  Bortezomib : the maximum tolerated dose (MTD) of bortezomib in combination with high-dose melphalan as a conditioning regimen for autologous stem cell transplant
  PBSCT : PBSCT #1 Day 0 PBSCT #2 Day 0 (approx 90 days =/- 15 days after PBSCT #1)
  Melphalan : Day -4 melphalan 100 mg/m2 intravenously over 30 minutes, Day -3 melphalan 100 mg/m2 intravenously over 30 minutes
Period: Overall Study
Arm/Group | Autologous PBSCT
Started | 30
Completed | 25
Not Completed | 5
Not completed — ineligible | 5

BASELINE CHARACTERISTICS:
Arm/Group | Autologous PBSCT
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Median overall survival after first peripheral blood stem cell transplant (PBSCT).
Time Frame: 40 months post transplant
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Autologous PBSCT
Number analyzed (Participants) | 25
months | 40 [32 to 40]

ADVERSE EVENTS:
Time Frame: 2 years post transplant
Arm/Group | Autologous PBSCT
Serious Adverse Events (participants affected / at risk) | 25/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous PBSCT (N=25)
Febrile Neutropenia (Infections and infestations) | 13
Bacteremia (Infections and infestations) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 7
Mucositis (Gastrointestinal disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2

LIMITATIONS AND CAVEATS:
per protocol subjects are followed for 2 years post transplant; however, subjects are followed on our long-term follow-up protocol(MCC12567/IRB6101) to assess overall and disease free survival. additional data available at time manuscript was written

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No